CLINICAL TRIAL: NCT05574647
Title: Evaluating the Role of Biparametric MRI and Image-fusion Targeted Biopsies for Detection of Prostate Cancer
Brief Title: Imperial Prostate 7 - Prostate Assessment Using Comparative Interventions - Fast Mri and Image-fusion for Cancer
Acronym: IP7-PACIFIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Cancer Research UK (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 22CX7488
Record Dates: First submitted 2022-08-03; First posted 2022-10-10 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer; Adenocarcinoma; Prostatic Neoplasms; Prostatic Diseases; Neoplasms
Keywords: Prostate Cancer; Prostate-Specific Antigen; bpMRI; mpMRI; Prostate biopsy; Multi-parametric MRI; Biparametric MRI
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma; Prostatic Diseases; Neoplasms

STUDY DESIGN:
Intervention Model Description: two linked RCTs which will test whether bpMRI and image-fusion make a difference if used in clinical practice, across multiple centres, without the incorporation bias inherent in paired-cohort studies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard: mpMRI (No Intervention): Participants will undergo mpMRI. Blinding will not be possible. Once the MRI report is issued, the local clinical team will make a decision about advising whether a biopsy is necessary or not.
- Intervention 1: bpMRI (Active Comparator): Participants will undergo bpMRI. Blinding will not be possible. Once the MRI report is issued, the local clinical team will make a decision about advising whether a biopsy is necessary or not.
  Interventions: Diagnostic Test: bpMRI
- Standard: Visual estimation targeted and systematic biopsy (No Intervention): Randomisation 2 will only be relevant if participants are advised by their clinical team to have a biopsy based on their MRI and other clinical factors. Participants advised to have a biopsy will undergo a visual estimation targeted biopsy
- Intervention 2: Image-fusion targeted and systematic biopsy (Active Comparator): Randomisation 2 will only be relevant if participants are advised by their clinical team to have a biopsy based on their MRI and other clinical factors. Participants advised to have a biopsy will undergo an image fusion targeted biopsy.
  Interventions: Diagnostic Test: Image-Fusion targeted and systematic Biopsy

INTERVENTIONS:
Diagnostic Test: bpMRI — biparametric MRI takes 30-40 minutes and requires a contrast injection called gadolinium (like a dye). This is also called long MRI and is most commonly used in the NHS.
  Other Names: biparametric MRI
  Arms: Intervention 1: bpMRI
Diagnostic Test: Image-Fusion targeted and systematic Biopsy — During image fusion targeted biopsy, the biopsy operator uses the MRI scans that were taken beforehand but laid on top of the live ultrasound images during the biopsy. This uses software and takes a few minutes longer to perform. Once the MRI images and ultrasound images are 'fused', the actual biopsies are taken as normal.
  Arms: Intervention 2: Image-fusion targeted and systematic biopsy

SUMMARY:
To evaluate the role of biparametric MRI and image-fusion targeted biopsies for the detection of prostate cancer.

To determine whether biparametric MRI (bpMRI) could be recommended as an alternative to multiparametric MRI (mpMRI) for the detection of clinically significant prostate cancers in patients at risk.

To determine whether image-fusion targeted biopsy is better than visual-registration (cognitive) targeted biopsy at detecting clinically significant prostate cancers in patients requiring prostate biopsy due to a suspicious MRI.

DETAILED DESCRIPTION:
Background and study aims:

The aim of this study is to improve the way prostate cancer is diagnosed by looking at two different types of MRI scans and two different types of prostate biopsy (tissue samples). A large study such as this is required to help the NHS decide how to diagnose prostate cancer in the future. If a person is suspected of having prostate cancer, then they are referred by their GP. At the hospital clinic, the participant will then have an MRI scan. If this scan shows that cancer might be present, then the doctor will usually suggest that the patient has a biopsy. There are two ways of doing a prostate MRI. One takes 30-40 minutes and requires a contrast injection called gadolinium (like a dye). This is called long MRI and is most commonly used in the NHS. Gadolinium is safe as it rarely causes any bad reaction but using it means that the scan takes more time. Another type of MRI takes 15-20 minutes and does not use gadolinium contrast. This is called a short MRI. Many studies over the last 5 years have shown that the long and short MRIs are similar in their accuracy in diagnosing important prostate cancer. These studies have not been of high quality or large enough to change NHS practice. Patients with suspicious areas on the MRI are usually advised to have a prostate biopsy. This involves taking tissue samples using a needle. The samples are then looked at under the microscope by a pathologist to see if cancer cells are present. There are two ways of doing a prostate biopsy. One is where the person doing the biopsy decides where to put the biopsy needle by looking at the MRI scans that have been already taken on a computer screen. The needle is guided to the prostate using live ultrasound scans that are shown on a different screen near the patient. The biopsy operator makes a judgement about where to place the biopsy needles. This is called visual registration. Tissue samples from other areas of the prostate that look normal on the MRI scans are also taken to ensure cancer is not missed. The other type of biopsy is called image fusion. During image fusion biopsy, the biopsy operator uses the MRI scans that have been taken beforehand but laid on top of the live ultrasound images during the biopsy. This uses software and takes a few minutes longer to perform. Once the MRI images and ultrasound images are 'fused', the actual biopsies are taken as normal. Studies over the last 5 years have shown mixed results. Some have shown that image fusion biopsy is no better than visual registration biopsy, whilst a few have shown it might make a difference in improving cancer detection. As a result, it is not known for certain which way is better. A large study is needed to show whether the investigators need to do image fusion or not, in order for the NHS to decide whether or not to use it in all hospitals doing prostate biopsies.

ELIGIBILITY:
Randomisation 1

Inclusion Criteria:

* Age 18 years or above (no upper limit)
* Patients with a prostate (either cis-male gender or trans-female gender with no prior androgen deprivation hormone use at all).
* Referred to hospital and advised to undergo a prostate MRI because of an abnormal digital rectal examination (regardless of PSA level) and/or an elevated PSA (within 6 months of screening visit) PSA >/=3.0ng/ml for age 50-69 years PSA >/=5.0ng/ml for age >/=70 years If family or ethnic risk for prostate cancer, PSA >/=2.5ng/ml for age 45-49 years

Exclusion Criteria:

* PSA >50ng/ml
* Prior prostate MRI or prostate biopsy in the two years prior to screening visit
* Prior diagnosis of prostate cancer
* Contraindication to MRI or gadolinium contrast
* Previous hip replacement to both hips
* Contraindication to performing a biopsy guided by a transrectal ultrasound probe

Randomisation 2

Inclusion Criteria:

* Visible suspicious finding on mpMRI or bpMRI from randomisation 1 requiring a targeted biopsy (MRI score 3, 4, 5 on either Likert or PIRADS schema)

Exclusion Criteria:

* As above for randomisation 1
* Patient refusal for biopsy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with a prostate (either cis-male gender or trans-female gender with no prior androgen deprivation hormone use at all)
Enrollment: 3600 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Randomisation 1: Proportion of clinically significant cancers detected in the randomised population of patients at risk. | maximum 12 weeks following enrolment
  Proportion of clinically significant cancers, defined as any amount of Gleason ≥3+4 (ISUP Grade Group ≥2) on biopsy, detected in the randomised population of patients at risk.
Randomisation 2: Proportion of clinically significant cancers detected in the randomised population of patients biopsied for a suspicious MRI. | maximum 12 weeks following enrolment
  Proportion of clinically significant cancers, defined as any amount of Gleason ≥3+4 (ISUP Grade Group ≥2) on biopsy, detected in the randomised population of patients biopsied for a suspicious MRI.

SECONDARY OUTCOMES:
MRI related adverse events | maximum 12 weeks following enrolment
  MRI related adverse events measured using documentation
MRI related serious adverse events | maximum 12 weeks following enrolment
  MRI related serious adverse events measured using documentation
Biopsy related adverse events | maximum 12 weeks following enrolment
  biopsy-related adverse events measured using documentation
Biopsy related serious adverse events | maximum 12 weeks following enrolment
  biopsy-related serious adverse events measured using documentation
The proportion of patients advised to undergo a needle biopsy after MRI | maximum 12 weeks following enrolment
  The proportion of patients advised to undergo a needle biopsy. The researchers will document common reasons for patients who are advised to undergo a biopsy or advised against a needle biopsy and still choose to have a biopsy.
The proportion of patients advised to undergo a prostrate biopsy after MRI | maximum 12 weeks following enrolment
  The proportion of patients undergoing a prostate biopsy after MRI. The researchers will document common reasons for patients who are advised to undergo prostrate biopsy after MRI.
The proportion of patients diagnosed with clinically significant prostates cancers on needle biopsy | maximum 12 weeks following enrolment
  The proportion of patients diagnosed with clinically significant prostates cancers defined as any Gleason 3+3=6 on needle biopsy carried out after MRI.
The proportion of patients diagnosed with clinically significant prostate cancers on prostate biopsy carried out after MRI | maximum 12 weeks following enrolment
  The proportion of patients diagnosed with clinically significant prostate cancers using other histological thresholds on prostate biopsy carried out after MRI.
  The researchers will evaluate these proportions by MRI score at patient and lesion level (on a scale of 1 to 5) and by the presence or absence of clinical risk parameters.
The proportion of patients diagnosed with clinically significant prostate cancers with targeted biopsy using four targeted cores | maximum 12 weeks following enrolment
  The proportion of patients diagnosed with clinically significant prostate cancers using all histological thresholds on targeted biopsy using four targeted cores
The proportion of patients diagnosed with clinically significant prostate cancers with targeted biopsy using six targeted cores | maximum 12 weeks following enrolment
  The proportion of patients diagnosed with clinically significant prostate cancers using all histological thresholds on targeted biopsy using six targeted cores
Detection rates for each randomised group of known prognostic risk categories | maximum 12 weeks following enrolment
  Detection rates for each randomised group of known prognostic risk categories. These are D' Amico, National Comprehensive Cancer Network (NCCN) and Cambridge Prognostic Groups (CPG).
Use Likert MRI scoring system to analyse the proportion of patients biopsied | maximum 12 weeks following enrolment
  A comparison of the two MRI scoring systems, Likert and PIRADS (the latest version as defined in MRI Reporting SOP), in terms of the proportion of patients biopsied and subsequently diagnosed with clinically significant and clinically insignificant prostate cancer, using each of the histological thresholds, on a prostate biopsy.
Use Prostate Imaging Reporting and Data System (PIRADS) MRI scoring system to analyse the proportion of patients biopsied | maximum 12 weeks following enrolment
  A comparison of the two MRI scoring systems, Likert and PIRADS (the latest version as defined in MRI Reporting SOP), in terms of the proportion of patients biopsied and subsequently diagnosed with clinically significant and clinically insignificant prostate cancer, using each of the histological thresholds, on a prostate biopsy.
Characteristics of cancer in targeted systematic biopsies | maximum 12 weeks following enrolment
  Characteristics of cancer in targeted versus systematic biopsies by MRI score, PSA, PSA density, age, ethnicity, family history and history of prior prostate biopsy with a multivariable evaluation to determine whether patients might avoid systematic sampling in the future.
Characteristics of cancer in targeted biopsies | maximum 12 weeks following enrolment
  Characteristics of cancer in targeted versus systematic biopsies by MRI score, PSA, PSA density, age, ethnicity, family history and history of prior prostate biopsy with a multivariable evaluation to determine whether patients might avoid systematic sampling in the future.
External validation of the Imperial Rapid Access to Prostate Imaging and Diagnosis (RAPID) Risk Score (MRI+) | maximum 12 weeks following enrolment
  External validation of the Imperial RAPID Risk Score (MRI+) within each randomised group of the IP7-PACIFIC study, external validation
External validation of the Imperial Rapid Access to Prostate Imaging and Diagnosis (RAPID) Risk Score in (Systematic+) | maximum 12 weeks following enrolment
  External validation of Imperial Rapid Access to Prostate Imaging and Diagnosis(RAPID) Risk Score (Systematic+) within each randomised group of the IP7-PACIFIC study, external validation
Impact of prostate biopsy in first randomised group (bpMRI) on patient-reported outcomes | maximum 12 weeks following enrolment
  Impact of prostate biopsy in each randomised group on patient-reported outcomes using a survey that includes EQ-5D-5L health-related quality of life questionnaire
Impact of prostate biopsy in second randomised group (mpMRI)on patient-reported outcomes | maximum 12 weeks following enrolment
  Impact of prostate biopsy in each randomised group on patient-reported outcomes using a survey that includes EQ-5D-5L health-related quality of life questionnaire
Impact of prostate biopsy in first randomised group (bpMRI) on patient-reported experience measures | maximum 12 weeks following enrolment
  Impact of prostate biopsy in each randomised group on patient-reported experience measures using version of the Prospective cohort study (Prostate Biopsy Effects: ProBE) questionnaire.
Impact of prostate biopsy in second randomised group (mpMRI) on patient-reported experience measures | maximum 12 weeks following enrolment
  Impact of prostate biopsy in each randomised group on patient-reported experience measures using version of the Prospective cohort study (Prostate Biopsy Effects: ProBE) questionnaire.
Analysis of biopsy rate in cancer detection (by all histological thresholds) during the time of study | maximum 12 weeks following enrolment
  Analysis of biopsy rates in cancer detection (by all histological thresholds) in the randomised group will be conducted by centre using centre size.
  MRI scanner type (1.5 Tesla vs. 3.0 Tesla), type of biopsy route used (transrectal vs trans perineal), number of systematic biopsies taken (limited systematic vs extended systematic biopsy), type of analgesia/anaesthetic (local anaesthetic, sedation or general anaesthetic) as additional stratification factors

CONTACTS AND LOCATIONS:
Locations (15):
- United Kingdom (15):
  - Southend University Hospital, Southend-on-Sea, Essex
  - University Hospital Southampton, Southampton, Hampshire
  - Medway Maritime Hospital, Gillingham, Kent
  - Basingstoke Hospital, Basingstoke
  - Southmead Hospital, Bristol
  - Addenbrooke Hospital, Cambridge, Cambridge
  - Cumberland Infirmary, Carlisle
  - St Peters Hospital, Chertsey
  - Darent valley Hospital, Dartford
  - Northwick Park Hospital, Harrow
  - St James's Hospital, Leeds, Leeds
  - Charing Cross Hospial, London
  - Manchester Royal Infirmary, Manchester
  - Northampton General Hospital, Northampton
  - Hillingdon Hospital, Uxbridge

IPD SHARING:
Plan to Share IPD: No